CLINICAL TRIAL: NCT04072861
Title: A Phase 1b Dose-escalating Study With RBT-9 in Healthy Volunteers and Volunteers With Chronic Kidney Disease Stage 3/4
Brief Title: A Study of RBT-9 in Healthy Volunteers and Volunteers With Stage 3/4 Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Renibus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: REN-003
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2023-12

CONDITIONS: Healthy Volunteers; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — tin protoporphyrin IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 9 mg (Experimental)
  Interventions: Drug: RBT-9
- 27 mg (Experimental)
  Interventions: Drug: RBT-9
- 90 mg (Experimental)
  Interventions: Drug: RBT-9

INTERVENTIONS:
Drug: RBT-9 — intravenous administration

SUMMARY:
This is a Phase 1b, single-center, dose-escalating study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamic effect of RBT-9 in healthy volunteers and in subjects with Stage 3/4 CKD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects age 18 to 80 years (inclusive, at time of ICF).
2. Body weight <125 kg.
3. Able and willing to comply with all study procedures.
4. Female subjects must be either post-menopausal for at least 1 year or surgically sterile (tubal ligation, hysterectomy or bilateral oophorectomy) for at least 3 months, or if of childbearing potential, have a negative pregnancy test and agree to use dual methods of contraception, or abstain from sexual activity from Screening until 28 days after study drug administration.

   Male subjects with female partners of childbearing potential must agree to use a highly effective method of contraception from screening until 28 days after study drug administration. All fertile men with female partners of childbearing potential should be instructed to contact the Investigator immediately if they suspect their partner might be pregnant (e.g., missed or late menstrual period) at any time during study participation.
5. CKD stage 3 as determined by a GFR between 30-59 ml/min as estimated using the CKD-EPI equation.
6. CKD stage 4 as determined by a GFR between 15-29 ml/min as estimated using the CKD-EPI equation.

Exclusion Criteria:

1. History of malignancy, except carcinoma in situ in the cervix, early stage prostate cancer or non-melanoma skin cancers. Cancer free for less than 5 years.
2. Use of investigational drugs or participation in another clinical trial within 30 days or 5 half-lives prior to Screening, whichever was longer.
3. Serum ferritin >500 ng/mL or received IV iron within 28 days of Screening.
4. Women who are pregnant, breastfeeding, or planning to become pregnant while participating in the study.
5. Any significant acute or chronic diseases, excluding CKD (≥ 15 ml/min); if CKD is present, those not at their baseline of renal function.
6. Abnormal Baseline liver tests or hepatitis serologies that suggest active infection.
7. Regular use of drugs of abuse and/or positive findings on urinary drug screening.
8. Current tobacco use and/or positive findings on urinary cotinine screening.
9. Severely physically or mentally incapacitated and who, in the opinion of Investigator, are unable to perform the subjects' tasks associated with the protocol.
10. Presence of any condition which, in the opinion of the Investigator, places the subject at undue risk or potentially jeopardizes the quality of the data to be generated.
11. History of photosensitivity or active skin disease which, in the opinion of the Investigator, could increase the risk of photosensitivity.
12. Known hypersensitivity or previous anaphylaxis to RBT-9 or tin-based product.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-03-31 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Riverside Clinical Research, Edgewater, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: It was pre-specified to analyze healthy volunteers and participants with CKD Stage 3/Stage 4 together and report results by dose.
Groups:
- 9 mg; 27 mg; 90 mg: Single IV infusion
Period: Overall Study
Arm/Group | 9 mg | 27 mg | 90 mg
Started | 6 | 18 | 18
Completed | 6 | 18 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 9 mg | 27 mg | 90 mg | Total
Number analyzed (Participants) | 6 | 18 | 18 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (11.69) | 59.3 (18.50) | 64.3 (15.29) | 59.5 (17.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 9 | 8 | 17
  Male | 6 | 9 | 10 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3 | 6
  Not Hispanic or Latino | 6 | 15 | 15 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 5 | 13
  White | 2 | 11 | 10 | 23
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3 | 6
Weight [Mean (Standard Deviation); unit: kg] | 92.6 (18.79) | 87.2 (16.84) | 88.6 (20.04) | 88.6 (18.18)
Height [Mean (Standard Deviation); unit: cm] | 175.9 (12) | 168.4 (10.11) | 170.3 (8.96) | 170.3 (9.97)
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.8 (3.87) | 30.8 (6.22) | 30.5 (6.71) | 30.5 (6.05)

OUTCOME MEASURES:

1. Primary Outcome: Effect of RBT-9 on Plasma Ferritin Levels
Description: Percent Change in Plasma Ferritin From Baseline to 24 hours
Time Frame: 24 hours post-infusion
Population: 1 value was missing at the 24 h timepoint from the 90 mg group
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | 9 mg | 27 mg | 90 mg
Number analyzed (Participants) | 6 | 18 | 17
Percent change from baseline | -9.83 [-34.22 to 14.56] | 7.66 [-6.41 to 21.73] | 39.37 [24.96 to 53.77]

2. Primary Outcome: Effect of RBT-9 on Plasma HO-1 Levels
Description: Percent Change in Plasma HO-1 From Baseline to 24 hours
Time Frame: 24 hours post-infusion
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | 9 mg | 27 mg | 90 mg
Number analyzed (Participants) | 6 | 18 | 18
Percent change from baseline | -16.07 [-68.78 to 36.65] | 10.46 [-19.66 to 40.58] | 33.37 [3.12 to 63.62]

3. Primary Outcome: Effect of RBT-9 on Plasma IL-10 Levels
Description: Percent Change in Plasma IL-10 From Baseline to 24 hours
Time Frame: 24 hours post-infusion
Population: Values at either baseline and/or the 24 h timepoint were missing from each of the treatment groups
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | 9 mg | 27 mg | 90 mg
Number analyzed (Participants) | 3 | 14 | 16
Percent change from baseline | 1.07 [-304.85 to 306.98] | 153.11 [10.49 to 295.73] | 752.53 [619.11 to 885.94]

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | 9 mg | 27 mg | 90 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 2/6 | 4/18 | 14/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 9 mg (N=6) | 27 mg (N=18) | 90 mg (N=18)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion Site Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection Site Bruising (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral Edema (General disorders) | 0 (0) | 1 (1) | 2 (2)
Ligament Sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 13 (13)
Contusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulum Intestinal Hemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Carboxyhaemoglobin Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT04072861/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-28): https://cdn.clinicaltrials.gov/large-docs/61/NCT04072861/SAP_001.pdf